CLINICAL TRIAL: NCT01461798
Title: Assessment of the Efficacy of Plant Stanol Esters in Reducing Cholesterol, Medellin 2011
Acronym: Ben2011
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jose María Maya Mejía (Other)
Responsible Party: Sponsor-Investigator, Jose María Maya Mejía, Johanna Romero Palacio, CES University
Organization: CES University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Ben2011
Record Dates: First submitted 2011-10-20; First posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Risk Reduction Behavior
Keywords: plant stanols; lipids; cardiovascular disease
MeSH Terms: conditions — Risk Reduction Behavior; Cardiovascular Diseases | interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benecol (Experimental): In 2009, the dairy Cooperative Colanta Launches Benecol ® yogurt, a product with optimal daily dose of plant stanol, each portion of 100 g containing 3.4 g of Benecol ®, corresponding to 2 g of plant stanol esters . Skim yogurt with Benecol ® is a product made from pasteurized skim milk, sweetened with sucralose homogenized and fermented by the action of specific lactic culture to obtain the optimal characteristics of texture and acidity. With the addition of fruit pulp and supplemented with plant stanol esters (Benecol ®) to help reduce the risk of cardiovascular disease (31). According to Weiss et al, drinkable yogurt with Benecol ® reduces total cholesterol by 5.8% and 9.8% in LDL cholesterol (32).
  Interventions: Dietary Supplement: assessment of efficacy of Benecol yogurt; Dietary Supplement: Placebo Yogurt
- yogurt (Placebo Comparator): Yogurt without plant stanols
  Interventions: Dietary Supplement: yogurt

INTERVENTIONS:
Dietary Supplement: assessment of efficacy of Benecol yogurt — Benecol Yogurt and Yogurt placebo for 4 weeks each, at a dose of 100 ml (200 ml in total) of yogurt twice a day with main meals
  Other Names: Benecol Yogurt; Placebo Yogurt
  Arms: Benecol
Dietary Supplement: Placebo Yogurt — Yogurt without the active principle
  Other Names: Colanta Yogurt
  Arms: Benecol
Dietary Supplement: yogurt — yogurt without plant stanols
  Other Names: Yogurt Colanta
  Arms: yogurt

SUMMARY:
Introduction:

Cardiovascular diseases have become the leading cause of death from chronic diseases in the world. One of the major risk factors for this disease is hypercholesterolemia, caused in most cases by a rich-fat diet, so came to our country Benecol ® yogurt, whose active ingredient is plant stanol ester that competes with total cholesterol and low density lipoprotein or LDL cholesterol by preventing them to be absorbed by the body and reducing blood levels.

Objective: To evaluate the efficacy of plant stanol ester in Benecol ® yogurt lowering blood lipids in moderately hypercholesterolemic patients treated at the CES Clinic during 2011.

Methods: A randomized crossover clinical trial, double-blind, placebo-controlled study in patients between 20 and 50 years with moderate hypercholesterolemia and are cared for CES control clinic in Medellin.

Expected results: Test the effectiveness of plant stanol esters in reducing total cholesterol and LDL cholesterol in patients with moderate hypercholesterolemia.

DETAILED DESCRIPTION:
The main cause of death worldwide are cardiovascular diseases, generated mainly by disturbances in the lipid profile. Several studies have shown that dyslipidemia is an important risk factor for this condition, thus maintaining the level of lipids in an appropriate range is ideal for preventing cardiovascular diseases (1)

Cardiovascular diseases are a serious epidemiological problem in the contemporary world, with approximately 17 million people die each year from causes such as myocardial infarction and stroke. The increase in cardiovascular disease and mortality attributable to them is a topic widely reported by several authors in the world. In Colombia after death from violent causes, cardiovascular diseases are on the second of the five leading causes of mortality in the general population.

Having high total cholesterol is a risk factor for the occurrence of various diseases of the circulatory system, therefore it is important to keep total cholesterol below 200 mg / dl and LDL cholesterol levels under 150 mg/dl, to avoid the accumulation of fat within the walls of the arteries that can lead to the formation of atherosclerotic plaques that cause decreased blood flow

The atlas published by WHO in 2005 provides comprehensive data on morbidity and mortality attributable to noncommunicable diseases, which are increasing. It is estimated that in 2001 approximately 60% of the 56.5 million deaths worldwide and 46% of diseases are due to noncommunicable diseases. The epidemiological burden of these diseases will increase to 57% by the year 2020. Almost 50% of deaths due to noncommunicable diseases are due to cardiovascular disease. By 2020, these diseases are responsible for 75% of all deaths worldwide.

Given the high prevalence of cardiovascular disease and dyslipidemia are considered a high risk factor for these occur, it is necessary to test the effectiveness of including the consumption of plant stanol esters in the diet to lower cholesterol values Total and LDL Cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Sign voluntarily the informed consent
* Male or female 20 to 50 years
* The concentration of total serum cholesterol of 5.2 - 7.5 mmol / l (205-290 mg / dl) at the screening visit (Visit 1 to 2 week)

Exclusion Criteria:

* Lipid-lowering medication or other drugs that significantly affect lipid values
* Diabetes Type I or II
* Severe obesity (BMI greater than 35 kg/m2)
* Fasting serum triglycerides> 4.0 mmol / l
* Liver or kidney disorder according to medical history
* History of coronary revascularization percutaneous transluminal coronary angioplasty within six months prior to screening
* History of temporary ischemic attack or stroke within six months prior to screening
* History of cancer or other malignant disease in the last five years
* Consumption of more than 15 parts of alcohol/week
* Pregnant or lactating
* Benecol consumption in your diet, or other plant sterol enriched products 30 days before visit 2 (Week 1), these will be identified by the survey
* Severe lactose intolerance, milk allergy or any other form of intolerance to the ingredients of the test products
* Celiac Disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Benecol Efficacy | 9 weeks
  Week 1: it will be taken a blood sample for lipid profile and other tests of liver and kidney function, patients will begin the Benecol ® yogurt consumption or placebo for four weeks, at week 5 it will be taken a new blood sample to perform mentioned test lipid levels and meet and determine the changes presented, patients will have a wash out week in Week 6 and groups will change for four weeks, at the end of week 9 will be held the last shot of sample for all tests again

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Romero, BML, Principal Investigator — CES University

REFERENCES:
- [Background] Furgione A y col. Dislipidemias primarias como factor de riesgo para enfermedad coronaria.Revista latinoamericana de hipertensión. 2009;4(1)
- [Background] Miettinen TA, Puska P, Gylling H, Vanhanen H, Vartiainen E. Reduction of serum cholesterol with sitostanol-ester margarine in a mildly hypercholesterolemic population. N Engl J Med. 1995 Nov 16;333(20):1308-12. doi: 10.1056/NEJM199511163332002. PMID 7566021
- [Background] Schmidt B, Ribnicky DM, Poulev A, Logendra S, Cefalu WT, Raskin I. A natural history of botanical therapeutics. Metabolism. 2008 Jul;57(7 Suppl 1):S3-9. doi: 10.1016/j.metabol.2008.03.001. PMID 18555851
- [Background] Katan et al. El efecto del éster estanol vegetal. Revista Europea de Nurición Clínica. 2009;63:2-10
- [Background] Musa-Veloso K et al. Una comparación entre la eficacia para disminuir el colesterol - LDL de los estanoles vegetales y los esteroles vegetales dentro de un rango de dosis continúo: Resultados de un meta-análisis de estudios controlados randomizados con placebo. 2011
- [Background] Plat J, van Onselen EN, van Heugten MM, Mensink RP. Effects on serum lipids, lipoproteins and fat soluble antioxidant concentrations of consumption frequency of margarines and shortenings enriched with plant stanol esters. Eur J Clin Nutr. 2000 Sep;54(9):671-7. doi: 10.1038/sj.ejcn.1601071. PMID 11002377
- [Result] Calvo Romero JM, Lima Rodriguez EM. ["Natural" treatments of hypercholesterolemia]. Rev Clin Esp. 2006 Nov;206(10):504-6. doi: 10.1157/13094900. Spanish. PMID 17129518
- [Result] Gylling H, Hallikainen M, Nissinen MJ, Miettinen TA. The effect of a very high daily plant stanol ester intake on serum lipids, carotenoids, and fat-soluble vitamins. Clin Nutr. 2010 Feb;29(1):112-8. doi: 10.1016/j.clnu.2009.08.005. Epub 2009 Aug 26. PMID 19709787
- [Derived] Vasquez-Trespalacios EM, Romero-Palacio J. Efficacy of yogurt drink with added plant stanol esters (Benecol(R), Colanta) in reducing total and LDL cholesterol in subjects with moderate hypercholesterolemia: a randomized placebo-controlled crossover trial NCT01461798. Lipids Health Dis. 2014 Aug 6;13:125. doi: 10.1186/1476-511X-13-125. PMID 25099071